CLINICAL TRIAL: NCT05727358
Title: Effectiveness of Group Acceptance and Commitment Therapy in Treating Acute Stroke Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PLA Rocket Force Characteristic Medical Center (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Liu Yun-e, Head nurse, PLA Rocket Force Characteristic Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z181100001718041
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-12

CONDITIONS: Acute Stroke Patients With Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): G-ACT
  Interventions: Behavioral: Group-based Acceptance and Commitment Therapy
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Group-based Acceptance and Commitment Therapy — G-ACT treatment in this study comprised 7 sessions of 45-60 minutes and was administered throughout the course of the 4-week long trial.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to discover the effectiveness of group-based Acceptance and Commitment Therapy (ACT) in treating depression for acute stroke patients. The main question[s] it aims to answer are:

* Group-based ACT (G-ACT) could significantly reduce the depressive symptoms in patients with acute stroke,
* the interventional efficacy could be maintained at 3-month follow-up
* similar benefits would be observed for quality of life (QOL), sleep quality, psychological flexibility, cognitive fusion, and confidence.

The patients included to the control group received usual care support in hospital, and the patients included to the intervention group received G-ACT and usual care support. the G-ACT treatment in this study comprised 7 sessions of 45-60 minutes and was administered throughout the course of the 4-week long trial.

ELIGIBILITY:
Inclusion Criteria:

1. primary diagnosis of acute stroke, the last onset occurred within 2 weeks
2. being over 18 years old
3. scoring at least 8 on the HAMD scale
4. Be conscious and able to communicate effectively with researchers
5. Primary school education level or above, 6) having signed informed consent.

Exclusion Criteria:

1. having a history of mental illness (such as bipolar disorder) or dementia, using psychiatric drugs or sedatives within 6 months, or currently using antidepressants
2. a diagnosis of cognitive impairment
3. receiving a psychological therapy in the previous three months, or currently experiencing severe psychotic symptoms
4. a history of drug abuse or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale (HAMD or HDRS, 24 item) | immediately after the intervention
  Each item is scored from 0 to 2 or 0 to 4, a higher score indicates much more serious depression
The Hamilton Depression Rating Scale (HAMD or HDRS, 24 item) | 3 months after the intervention
  Each item is scored from 0 to 2 or 0 to 4, a higher score indicates much more serious depression

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | immediately after and 3 months after the intervention
  physical component summary (PCS) and mental component summary (MCS) ranging from 0 (worst) to 100 (best).A higher score reflects better HRQoL
The Acceptance and Action Questionnaire II (AAQ-II) | immediately after and 3 months after the intervention
  the total score ranges from 7 to 49 with a higher score indicating less psychological flexibility.
The Cognitive Fusion Questionnaire (CFQ) | immediately after and 3 months after the intervention
  scores range from 0 to 63 with a higher score indicating more fused one is with one's thoughts
The confidence was assessed using the Confidence after Stroke Measure (CaSM) | immediately after and 3 months after the intervention
  total scores ranging from 0 to 81 and higher scores representing higher confidence.
The Pittsburgh Sleep Quality Index (PSQI) | immediately after and 3 months after the intervention
  total scores ranging from 0 to 21 and higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- The PLA Rocket Force Characteristic Medical Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu YE, Lv J, Sun FZ, Liang JJ, Zhang YY, Chen J, Jiang WJ. Effectiveness of group acceptance and commitment therapy in treating depression for acute stroke patients. Brain Behav. 2023 Dec;13(12):e3260. doi: 10.1002/brb3.3260. Epub 2023 Nov 8. PMID 37938871